CLINICAL TRIAL: NCT06418308
Title: Comparison of Intrathecal Epinephrine Versus Dexmedetomidine as Adjuvants in Cesarean Section
Brief Title: Intrathecal Dexmedetomidine vs Epinephrine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Vice Chair of Education Department of Anesthesiology, Pain, & Perioperative Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-23-01613
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section; Anesthesia, Spinal
Keywords: Cesarean Section; Spinal Anesthesia; Intrathecal adjuncts; Dexmedetomidine; Epinephrine
MeSH Terms: interventions — Dexmedetomidine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receiving the addition of epinephrine or dexmedetomidine to the standard spinal medication mixture of 10.25 mg hyperbaric bupivacaine, and 0.125 mg morphine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be assigned a group by picking from a stack of envelopes. The interventional drug which the envelope contains will be assigned by a random number generator. The interventional drug will be drawn up by an anesthesiologist not involved in the patient's care and the syringe given to the anesthesiologist performing the spinal anesthetic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): receiving the addition of 5 mcg of dexmedetomidine to the standard spinal medication mixture.
  Interventions: Drug: Dexmedetomidine; Drug: Standardized Spinal Mixture
- Epinephrine (Active Comparator): receiving the addition of 200 mcg of epinephrine to the standard spinal medication mixture
  Interventions: Drug: Epinephrine; Drug: Standardized Spinal Mixture

INTERVENTIONS:
Drug: Dexmedetomidine — 5 mcg of dexmedetomidine
  Arms: Dexmedetomidine
Drug: Epinephrine — 200 mcg of epinephrine
  Arms: Epinephrine
Drug: Standardized Spinal Mixture — Standardized spinal mixture of 10.25 mg hyperbaric bupivacaine, and 0.125 mg morphine.

SUMMARY:
Several studies have shown that adding dexmedetomidine or epinephrine to single-dose spinal analgesia preparations improves the length and/or speed of onset of the sensory block and post-operative pain management without increased negative side effects. To date, however, no study has compared adjunctive intrathecal dexmedetomidine to adjunctive intrathecal epinephrine in single-dose spinal analgesia. The purpose of this study is to determine if adjunctive intrathecal dexmedetomidine is non-inferior to adjunctive intrathecal epinephrine in providing better single-dose spinal analgesia during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients
* aged 18-55 years
* presenting for scheduled primary or secondary cesarean section
* candidates for single shot spinal anesthesia singleton pregnancy

Exclusion Criteria:

* patient refusal of spinal anesthetic
* if patient is not a candidate for spinal anesthesia due to history of coagulopathy, elevated intracranial pressure, infection at site of injection, etc.
* emergency cesarean section
* preexisting motor or sensory deficit
* suspected pre-eclampsia
* patient receiving combined spinal-epidural as anesthetic technique
* BMI > 40

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time required for sensory recovery | 270 minutes
  Investigate the efficacy of intrathecal epinephrine versus dexmedetomidine as adjuvant agents in cesarean section. Once the sensory block to pinprick has receded to a T10 level, the spinal is no longer as effective for surgical level pain relief. This is a measure of the duration of the spinal as an effective analgesic. Sensory recovery will be a T10 level. This will be measured in minutes.

SECONDARY OUTCOMES:
Time to Bromage Score 1 | 270 minutes
  Time to motor recovery determines how long the patient will be in the post anesthesia care unit. This will be measured in minutes. Bromage Scale to determine recovery where recovery will be Bromage 1.
  Bromage Scale:
  Bromage 0 full flexion knees and feet
  Bromage 1 just able to move knees
  Bromage 2 able to move feet only
  Bromage 3 unable to move feet or knees
Blood Pressure | 30 minutes
  Systolic and Diastolic Blood pressures will be measured preoperatively and then every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement.
Phenylephrine Infusion Rate | 2 to 30 minutes
  the phenylephrine infusion rate from 2 to 30 minutes after spinal placement
Total Phenylephrine Infusion | during surgery which can go up to 150 minutes
  the total phenylephrine infusion given during surgery.
Number of Phenylephrine Boluses | during surgery which can go up to 150 minutes
  Number of Phenylephrine Boluses given during the operation
Number of Ephedrine Boluses | during surgery which can go up to 150 minutes
  Number of Ephedrine Boluses given during the operation
Number of Nausea episodes | 60 minutes
  Nausea will be assessed every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement. If patient self-reports or exhibits any of these symptoms after 30 minutes while still in OR, this will also be recorded until patient is in PACU.
Number of Vomiting episodes | 60 minutes
  Vomiting will be assessed every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement. If patient self-reports or exhibits any of these symptoms after 30 minutes while still in OR, this will also be recorded until patient is in PACU.
Number of Shivering episodes | 60 minutes
  Shivering will be assessed every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement. If patient self-reports or exhibits any of these symptoms after 30 minutes while still in OR, this will also be recorded until patient is in PACU.
Number of Pruritus episodes | 60 minutes
  Pruritus will be assessed every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement. If patient self-reports or exhibits any of these symptoms after 30 minutes while still in OR, this will also be recorded until patient is in PACU.
Pain Score at Skin Incision | within the surgery, which can go up to 150 minutes
  Pain scores at time of skin incision. Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Pain Score at Uterine Incision | within the surgery, which can go up to 150 minutes
  Pain scores at time of uterine incision. Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Pain Score at Uterine Exteriorization | within the surgery, which can go up to 150 minutes
  Pain scores at time of uterine exteriorization. Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Pain Score at Uterine Closure | within the surgery, which can go up to 150 minutes
  Pain scores at time of uterine closure. Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Pain Score at Gutter Cleaning | within the surgery, which can go up to 150 minutes
  Pain scores at time of gutter cleaning. Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Pain Score at Procedure Finish | at procedure finish, which can go up to 150 minutes
  Pain scores at time of procedure finish . Pain will be graded on a scale of 0-10 (0 being no pain and 10 being the worst pain imaginable).
Additional IV Medication | during surgery which can go up to 150 minutes
  Any additional IV medications that need to be given during the surgery will be recorded (e.g. IV fentanyl).
Number of participants who require Conversion to General Anesthesia | during surgery which can go up to 150 minutes
  Number of participants who require Conversion to General Anesthesia. If converted to general anesthesia, enrollment in study will end.
Heart Rate | total of 30 minutes from the time of spinal placement.
  Heart rate will be measured every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement.
Oxygen Saturation | total of 30 minutes from the time of spinal placement.
  Oxygen saturation will be measured every 2 minutes for 10 minutes then every 5 minutes for a total of 30 minutes from the time of spinal placement.
Apgar Scores | 1 minute and 5 minutes
  Neonatal Apgar Scores at 1 and 5 minutes will be recorded. Apgar score ranges from 0 to 10, with higher score indicating better health outcomes.
Number of NICU admission | Day 1
  Number of babies that require Neonatal Intensive Care Unit (NICU) admission from the OR.
Patient Satisfaction Score | Post-Op Day 1
  Patient will be asked to score satisfaction postoperatively Patient Satisfaction Score
  1. Completely dissatisfied
  2. Partially dissatisfied
  3. Neutral
  4. Partially satisfied
  5. Completely satisfied
Time to First opioid | 24 hours
  Via chart review, time to first opioid within a 24 hour time period after spinal placement.
Total Opioid Dose | 24 hours
  Via chart review, time to total opioids given within a 24 hour time period after spinal placement.
Time to sensory block | 20 minutes
  Spinal Onset - The T4 sensory level is considered adequate for operative analgesia for cesarean delivery. Time to a sensory block to pinprick to T4 level over a 20 minute time period after spinal placement will be recorded. If T4 not reached, highest level achieved will be recorded. This will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan in place to share IPD.